CLINICAL TRIAL: NCT02085395
Title: An Open Phase II Study to Assess the Efficacy and Safety of Topical SR-T100® Gel in the Treatment of Human Cutaneous Squamous Cell Carcinoma in Situ (Actinic Keratosis and Bowen's Disease)
Brief Title: Clinical Study Assessment of SR-T100 Topical Gel Against Actinic Keratosis
Acronym: AK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCCD06003A
Record Dates: First submitted 2014-03-11; First posted 2014-03-12 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Actinic Keratosis; Bowen's Disease
Keywords: Actinic Keratosis, AK, Bowen's Disease, Bowen
MeSH Terms: conditions — Keratosis, Actinic; Bowen's Disease | interventions — SR-T100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SR-T100 ® Gel (Experimental): Topical gel containing 2.3% of solamargine in Solanum undatum extract is used once daily with occlusive dressing for 16 weeks.
  Interventions: Drug: SR-T100 ® Gel

INTERVENTIONS:
Drug: SR-T100 ® Gel
  Other Names: SR-T100

SUMMARY:
To evaluate the efficacy of SR-T100 gel by observing the lesion size (length x width x height) of human cutaneous squamous cell carcinoma in situ (Actinic Keratosis and Bowen's Disease) reduced at least 75%.

DETAILED DESCRIPTION:
An open phase II study to assess the efficacy and safety of topical SR-T100 gel in the treatment of human cutaneous cell carcinoma in situ (Actinic Keratosis and Bowen's Disease). The primary efficacy endpoint defines as the proportion of patients whose lesion size reduced at least 75%. The secondary efficacy endpoints include complete clearance rate as the proportion of patients with no clinical visible AK/BD lesions in the treatment area, partial clearance rate as the proportion of patients at least a 75% reduction of AK/BD lesion size in teh treatment area, and histological response rate as the proportion of patients with biopsy proven clearance of AK and BD in situ. Safety was evaluated by clinically significant changes occurring from baseline to the end of the study by observing physical examination, vital signs, laboratory assessments and AEs.

ELIGIBILITY:
Inclusion Criteria:

* Patients met ALL of the inclusion criteria for the entry of this study:

  1. Male or female; aged ≧ 20 years old.
  2. Patients had histologically confirmed Squamous cell carcinoma in situ (AK or BD) for the targeted lesion.
  3. Patients had a measurable lesion 5mm or larger for AK or 10mm or larger for BD.
  4. Patient had a performance status of < 2 (ECOG).
  5. Patients who had signed an approved written informed consent.

Exclusion Criteria:

* Patients were excluded from this study for ANY of the following reasons:

  1. Patients with histologic subtypes other than squamous cell carcinoma in situ (AK or BD).
  2. Patients with tumor extending into the oral cavity, nostrils, eyelids, urethra, anus, vagina or rectum.
  3. Patients who had grossly suspicious or inflamed nodes on physical examination.
  4. Patients with grossly infected tumors.
  5. Patients with recurrent invasive squamous cell carcinoma.
  6. Patients with a history of other invasive malignancies, if there was any evidence of the other malignancy being present within the past 5 years. Patients were also excluded if their previous cancer treatment contraindicated this protocol therapy.
  7. Use of any investigational drug in the 30 days before screening.
  8. Pregnant or lactating women or women of childbearing potential using inadequate contraceptive methods.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Partial clearance rate | 16 weeks treatment and 4 weeks follow-up
  To assess the response rate of SR-T100® gel in patients with cutaneous squamous cell carcinoma in situ (Actinic Keratosis: AK; and Bowen's Disease: BD), defined as the proportion of patients whose lesion size (length x width x height) reduced > 75%.

SECONDARY OUTCOMES:
Complete clearance rate | 16 weeks treatment and 4 weeks follow-up
Partial clearance rate | 16 weeks treatment and 4 weeks follow-up

OTHER OUTCOMES:
Histological response rate | 2-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hamm-Ming Sheu, MD, Principal Investigator — Department of Dermatology National Cheng Kung University Hospital Tainan, Taiwan, ROC
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan